CLINICAL TRIAL: NCT05075265
Title: Pharmacokinetics of Methadone in Adults Undergoing Cardiac Surgery With Extracorporeal Circulation
Brief Title: Methadone in Adults Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 200323005
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2021-09

CONDITIONS: Cardiosurgery; Cardiopulmonary Bypass; Methadone
Keywords: extracorporeal circulation; pharmakinetics
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Methadone Group: adult patients undergoing cardiac surgery with extracorporeal circulation
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — Standard dose of 0.2 ug/kg before Cardiopulmonary Bypass.

SUMMARY:
In cardiac surgery, the establishment of Cardiopulmonary bypass (CPB) involves profound changes that can alter the pharmacokinetics and clinical response to drugs. Methadone has characteristics that make it attractive for the management of postoperative pain, however, to date there are no pharmacokinetic or pharmacodynamic studies that allow guidance on how to perform the dosage and dose adjustment of methadone in patients undergoing cardiopulmonary bypass.

The main of this study is to describe the pharmacokinetics of methadone in adult patients undergoing cardiac surgery with extracorporeal circulation.

A pharmacokinetic clinical study will be proposed. Drug concentrations will be measured at different times, estimating how plasma levels vary before, during and after CPB. For the plasma methadone analysis, 10 blood samples will be taken from each patient following a pre-established schedule. They will be analyzed using a high performance liquid chromatography (HPLC) spectrofluorometric method.

Changes in volumes, clearance, and other covariates associated with CPB are not expected to significantly affect methadone plasma concentrations.

DETAILED DESCRIPTION:
Introduction:

Pharmacokinetics studies the processes of absorption, distribution, metabolism and excretion of a drug. There are multiple conditions that can affect the expected pharmacokinetic behavior of a drug. In cardiac surgery, for example, most surgeries require stopping the heart. For this, different cardioplegia solutions and an extracorporeal circulation machine (ECC) are used to allow oxygenation and blood circulation to continue to the rest of the body. The establishment of Cardiopulmonary bypass (CPB) involves profound changes that can alter the pharmacokinetics and clinical response to drugs. An adequate knowledge of the magnitude and direction of these changes is therefore necessary for each drug in particular, in order to achieve an optimal dosage at the time of use. In order to optimize postoperative pain management in cardiac surgery, other drugs have been used as an alternative to the usual management of boluses of morphine or fentanyl. Methadone has pharmacokinetic and pharmacodynamic characteristics that make it attractive; however, despite being a relatively old drug, its use in cardiac surgery is relatively recent. To date, few studies have been published with the use of methadone in a single intraoperative bolus scheme, both studies report positive results. However, to date there are no pharmacokinetic or pharmacodynamic studies that provide guidance on how to dose and adjust the dose of methadone in patients undergoing cardiopulmonary bypass in this context.

THEORETICAL FRAMEWORK Pharmacokinetics is the branch of pharmacology that studies the relationship between the dose of a drug and its plasma concentrations, "what the body does to the drug." Pharmacokinetics studies the processes of absorption, distribution, metabolism and excretion of a drug.

Compartment pharmacokinetic models emerge as a way of conceptualizing this study. They describe the organism as a set of compartments where each one represents a part of the biological material in which the drug is supposed to be uniformly distributed and has the same kinetic properties. It is possible to use 1 or more compartments to describe the kinetics of a drug. For the estimation of population parameters, specific study methods are required that allow the most accurate and precise estimation of population parameters, both of fixed effect, as well as of inter and intra-individual random effect. Among the available parametric methods, which assume a known probability distribution, one widely used is the non-linear mixed effects model. Proposed by Sheiner and Beal, it is currently the reference method in pharmacokinetic analysis in large population groups. This method allows estimating inter individual variability without ignoring the large number of limitations present in observational data.

From a clinical perspective, there are multiple conditions that can alter the expected pharmacokinetic behavior of a drug; diseases, for example, can modify the physiological functions of different organs, alter blood flow and alter the metabolism and elimination of some drugs. Another example is the case of cardiac surgery where, for the realization of most of the surgeries it is required to stop the heart. For this, different cardioplegia solutions and an extracorporeal circulation machine (CPB) are used to allow oxygenation and blood circulation to continue to the rest of the body during the surgical procedure. The establishment of CPB involves profound changes that can alter the pharmacokinetics and clinical response to drugs. An adequate knowledge of the magnitude and direction of these changes is therefore necessary for each drug in particular, in order to achieve an optimal dosage at the time of use.

At the start of CPB, acute hemodilution can cause a decrease in the plasma concentration of almost any drug. Hypothermia, frequently used in cardiac surgery, can also reduce metabolic activity in the liver and thus decrease metabolic clearance. The oxygenator membrane, reservoir filters, and ECC circuit can sequester varying amounts of some drugs. This occurs with fentanyl, for which a 25% decrease in plasma concentration upon entering CPB was initially described. A similar effect was described for sulfentanil. In the case of remifentanil that is metabolized by plasma esterases, a decrease in clearance is observed with hypothermia (6.3% per 1ºC). In this context, it has not been described how the pharmacokinetics of methadone could change in these patients.

Methadone is a synthetic opioid that has pharmacokinetic and pharmacodynamic characteristics that make it attractive for its perioperative use, both in acute pain and in chronic pain. Its long half-life allows more stable inter-dose plasma levels. Administered in a single dose of 0.2 to 0.3 mg / kg, it has not been associated with a higher incidence of adverse effects (compared to short-acting opioids), reaching a duration of analgesia between 24 hours and 35 hours. It is highly bound to plasma proteins. Between 60 and 90% circulates bound to proteins, mainly acid glycoprotein. Unlike morphine, it does not generate active metabolites after its liver biotransformation and does not accumulate in kidney failure, which allows its use in patients with chronic kidney disease or hemodialysis. It is inexpensive compared to other opioids. In addition to its action on opioid receptors, it reduces the re-uptake of serotonin and norepinephrine involved in acute and chronic pain processes. It also exerts antagonistic activity at NMDA glutamatergic receptors. Glutamate is the main excitatory amino acid of the central nervous system and participates in the processes of nociceptive transmission at the spinal level. Its action on pain pathways is mainly mediated through ionotropic receptors (AMPA, NMDA and Kainic) involved in the generation and maintenance of states of hyperalgesia (exacerbated response to noxious stimulus) and allodynia (decreased pain threshold). These properties give it potential effectiveness in relieving neuropathic pain, also showing good results in the treatment of chronic pain and cancer pain.

Adequate control of postoperative pain is a relevant issue in cardiac surgery. Poorly treated acute pain can produce serious deleterious effects, namely; activation of the sympathetic system, tachycardia, arrhythmias and ischemia due to increased myocardial oxygen consumption. Pulmonary adverse effects (atelectasis and pneumonia), gastrointestinal (ileus), musculoskeletal (muscle weakness), endocrine (hypoglycemia) and psychological (depression). The presence of these complications delays and makes recovery difficult. With current techniques, incidences of acute pain between 30 and 75% are reported, with greater intensity during the first 2 days. Patients with high levels of postoperative pain have 3.5 times the risk of chronic pain and their inadequate treatment can lead to chronic or neuropathic pain that is difficult to manage . The incidence of chronic pain after cardiac surgery can reach up to 30-40% of patients during the first year.

In this scenario, the methadone use could confer certain advantages. Its long half-life would allow the establishment of simplified dosage schedules with less variability in plasma levels between doses than with the usual management that considers fentanyl or morphine in intermittent boluses. Its pharmacokinetics allow its administration in one dose per day, regardless of the need and cost of a continuous infusion pump. Methadone could reduce the incidence of chronic pain by optimizing acute pain control and its anti-NMDA activity. Finally, cardioprotective properties have been described.

Despite being a relatively old drug, the use of methadone as an alternative to short-acting opioids (fentanyl or morphine) in cardiac surgery is relatively recent. Few studies have been published with the use of intraoperative methadone in cardiac surgery and two report an adequate clinical effect with positive results. Although the presence of an adequate postoperative clinical effect suggests that exposure to cardiac surgery with cardiopulmonary bypass alone does not produce a significant change in postoperative methadone concentrations, the actual pharmacokinetic behavior of methadone in these circumstances is unknown. To date, there are no pharmacokinetic or pharmacodynamic studies that provide guidance on how to dose and adjust the dose of methadone in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 45 and 75 years old who undergo surgery of coronary bypass with CPB, univalvular replacement, bivalvular or coronary bypass plus univalvular on a scheduled basis at the UC-Christus Clinical Hospital (HCUC) and that have ASA II-III classification.

Exclusion Criteria:

* BMI> 35, history of chronic liver damage, kidney damage with estimated creatinine clearance <60 ml / min, severe ventricular dysfunction (EF <30% or severe dysfunction in ventriculography), recent cerebrovascular accident (CVA) or sequelae, endocarditis, use of intraoperative ultrafiltration or methadone in the previous 36 hours.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients who undergo cardiac surgery whith cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Time Frame: 0, 5-10, 30, 60, 120, 240 minutes of operation of the CPB and 12 or 24 hours of CPB]
  Calculate maximum plasma concentration (Cmax) Methadone plasma levels measured with high pressure fluid (HPLC) after a single bolus of Methadone in enrolled adult Adults Undergoing Cardiac Surgery With Extracorporeal Circulation
Describe the change of the levels of methadone plasmatic levels (ng/mL) measured by high pressure liquid chromatography (HPLC) | Time Frame: 0, 5-10, 30, 60, 120, 240 minutes of operation of the CPB and 12 or 24 hours of CPB]
  Change of the plasmatic levels of Methadone [ Time Frame: The concentrations will be measured in time: 0, 5-10, 30, 60, 120, 240 minutes of operation of the CPB and 12 or 24 hours of CPB]

CONTACTS AND LOCATIONS:
Overall Officials: Wilbaldo Salas, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clinico Universidad Catolica, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mets B. The pharmacokinetics of anesthetic drugs and adjuvants during cardiopulmonary bypass. Acta Anaesthesiol Scand. 2000 Mar;44(3):261-73. doi: 10.1034/j.1399-6576.2000.440308.x. PMID 10714838
- [Background] Starkey ES, Sammons HM. Practical pharmacokinetics: what do you really need to know? Arch Dis Child Educ Pract Ed. 2015 Feb;100(1):37-43. doi: 10.1136/archdischild-2013-304555. Epub 2014 Aug 13. PMID 25122157
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Shear T, Parikh KN, Patel SS, Gupta DK. Intraoperative Methadone for the Prevention of Postoperative Pain: A Randomized, Double-blinded Clinical Trial in Cardiac Surgical Patients. Anesthesiology. 2015 May;122(5):1112-22. doi: 10.1097/ALN.0000000000000633. PMID 25837528
- [Derived] Salas WE, Cortinez LI, Lopez RA, Rolle A, Elgueta F, Godoy CO, Giordano A, Contreras V, Anderson BJ. Pharmacokinetics of Methadone in Adult Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass. Anesth Analg. 2025 Aug 1;141(2):384-392. doi: 10.1213/ANE.0000000000007312. Epub 2024 Nov 21. PMID 39773745